CLINICAL TRIAL: NCT02076165
Title: A Patient-Focused Approach to Insomnia Treatment for Women Veterans
Brief Title: Insomnia Treatment for Women Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIR 13-058
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Insomnia
Keywords: insomnia; women
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABC-I (Experimental): Participants completed a 5 session intervention, Acceptance and the Behavioral Changes to Treat Insomnia (ABC-I). This was considered the "new treatment" being studied.
  Interventions: Behavioral: Acceptance and the Behavioral Changes to Treat Insomnia
- CBT-I (Active Comparator): Participants received a 5-session intervention, cognitive-behavioral therapy for insomnia (CBT-I). This was considered the "standard care" treatment.
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia

INTERVENTIONS:
Behavioral: Acceptance and the Behavioral Changes to Treat Insomnia — Participants attended 5 individual sessions incorporating behavioral treatment components plus acceptance and commitment therapy (ACT) with a trained instructor.
  Other Names: ABC-I
  Arms: ABC-I
Behavioral: Cognitive behavioral therapy for insomnia — Participants attended 5 individual sessions incorporating behavioral and cognitive therapy components with a trained instructor.
  Other Names: CBT-I
  Arms: CBT-I

SUMMARY:
Women Veterans have high rates of insomnia. Prior research and our preliminary findings show that insomnia impacts the health and quality of life of women Veterans and that those with insomnia prefer non-medication treatments over sleeping pills. This study compared two non-medication behavioral treatments for insomnia to determine impacts on adherence rates and sleep/wake patterns. A novel treatment, Acceptance and the Behavioral Changes to Treat Insomnia (ABC-I) was compared to standard treatment, Cognitive Behavioral Therapy for Insomnia (CBT-I). The results showed that ABC-I was non-inferior to CBT-I and adherence to the treatments was similar in both groups. These results improve the repertoire of available behavioral treatments for insomnia within VA by showing that a new treatment, called ABC-I, works as well as standard CBT-I.

DETAILED DESCRIPTION:
The number of women Veterans is increasing due to changes in the composition of the active duty military, and understanding the healthcare needs of this growing segment of the patients we serve is critical. Insomnia complaints are more common among women than men, with a mean prevalence of over 23% among US women. Insomnia (defined as sleep disturbance that is sufficiently severe to cause distress or impact functioning), is a significant public health concern that contributes to lost productivity, psychological distress, medical morbidity, and mortality risk. In a recent paper on transformation of care for women Veterans, Yano et al. included "sleep issues" as part of the "VA Women's Health Research Agenda for the Future"; however, systematic reviews of VA women's health research (2006 and 2011) did not identify any prior studies of sleep disorders among women Veterans. In 2011 the investigators completed the first descriptive study of sleep problems among women Veterans who receive VA Healthcare (HSRD PPO 09-282-1; PI: Martin). The investigators found high rates of insomnia (54% of respondents) and comorbid conditions that may impact treatment acceptability and delivery. The investigators also found that women Veterans with insomnia preferred non-medication treatments over medications, and that they were most likely to access this treatment if it were delivered in individual format (rather than groups). There is a growing literature on treatment of insomnia among individuals with comorbid conditions, suggesting that insomnia treatment may lead to meaningful and durable improvements in sleep quality and other symptoms.

This study was a randomized trial to compare two non-medication behavioral treatments for insomnia. The first is a novel intervention based on Acceptance and Commitment Therapy (ACT) in addition to sleep restriction, stimulus control and sleep hygiene. this treatment is called Acceptance and the Behavioral Changes to Treat Insomnia (ABC-I). The standard treatment used as a comparator was Cognitive-Behavioral Therapy for Insomnia (CBT-I). The objectives were: 1) to compare dropout rates and adherence to behavioral recommendations between the two treatment programs, 2) to compare the effectiveness of the two treatment programs in improving sleep/wake patterns from baseline to post-treatment, and 3) to compare the maintenance of improvements in sleep/wake patterns across the two treatment programs 3-months after the end of treatment.

A brief survey was mailed to women Veterans who received healthcare within 6 months from the VA Greater Los Angeles Healthcare System, and women referred for treatment of sleep disorders were also invited to participate. All women who return the survey indicating symptoms of insomnia were contacted by phone and invited to participate in the treatment study. Exclusion criteria were limited to severe or unstable medical/psychiatric disorders, the presence of moderate-to-severe sleep apnea, or barriers to attending the treatment sessions (e.g., live too far away, no access to transportation). The insomnia treatment programs were provided in 5 one-on-one sessions to women Veterans with insomnia by a trained interventionist. Women Veterans will be randomized to one of the two treatment programs (ABC-I: n=74 and CBT-I: n=75). Adherence and attrition were measured in both treatment groups. Sleep quality (self-reported and objectively measured), psychiatric symptom severity and quality of life will be assessed at baseline, post-treatment and at 3-month follow-up. ANOVA was used to test for differences between groups in adherence and attrition. Equivalency/noninferiority methods were used to determine whether sleep-related outcomes are comparable between the two groups, using both intent to treat and per protocol analyses. A priori power calculations showed that there was sufficient power to identify clinically meaningful differences with 148 randomized participants.

ELIGIBILITY:
Inclusion Criteria:

* Female Veteran
* Community-dwelling
* Age 18 years and older
* Received care from VA Greater Los Angeles Healthcare System in the past six months
* Responses to postal survey indicate symptoms of insomnia
* Did not check "opt-out" box for further contact on postal survey
* Live within 50 mile radius of Sepulveda VA Ambulatory Care Center

Exclusion Criteria:

* Unstable housing
* No transportation to the medical center
* Current pregnancy
* Significant health or emotional problems, or use of drugs or alcohol
* Untreated sleep apnea
* Restless legs syndrome that accounts for the sleep disturbances reported
* Circadian rhythm sleep disorder that accounts for the sleep disturbances reported
* Active substance users or in recovery with less than 90 days of sobriety
* Unstable medical or psychiatric disorders (which is a contraindication for behavioral treatment of insomnia)
* Remission of insomnia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 347 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Martin, PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fung CH, Martin JL, Hays RD, Rodriguez JC, Igodan U, Jouldjian S, Dzierzewski JM, Kramer BJ, Josephson K, Alessi C. Development of the Usability of Sleep Apnea Equipment-Positive Airway Pressure (USE-PAP) questionnaire. Sleep Med. 2015 May;16(5):645-51. doi: 10.1016/j.sleep.2015.01.019. Epub 2015 Feb 12. PMID 25890783
- [Result] Dzierzewski JM, Mitchell M, Rodriguez JC, Fung CH, Jouldjian S, Alessi CA, Martin JL. Patterns and predictors of sleep quality before, during, and after hospitalization in older adults. J Clin Sleep Med. 2015 Jan 15;11(1):45-51. doi: 10.5664/jcsm.4362. PMID 25325580
- [Result] Culver NC, Song Y, Kate McGowan S, Fung CH, Mitchell MN, Rodriguez JC, Dzierzewski JM, Josephson KR, Jouldjian S, Washington DL, Yano EM, Schweizer CA, Alessi CA, Martin JL. Acceptability of Medication and Nonmedication Treatment for Insomnia Among Female Veterans: Effects of Age, Insomnia Severity, and Psychiatric Symptoms. Clin Ther. 2016 Nov;38(11):2373-2385. doi: 10.1016/j.clinthera.2016.09.019. Epub 2016 Oct 27. PMID 28314434
- [Result] Song Y, Washington DL, Yano EM, McCurry SM, Fung CH, Dzierzewski JM, Rodriguez JC, Jouldjian S, Mitchell MN, Alessi CA, Martin JL. Caregiving-Related Sleep Problems and Their Relationship to Mental Health and Daytime Function in Female Veterans. Behav Sleep Med. 2018 Jul-Aug;16(4):371-379. doi: 10.1080/15402002.2016.1228640. Epub 2016 Oct 3. PMID 27690634
- [Derived] Saldana KS, Carlson GC, Revolorio K, Kelly MR, Josephson KR, Mitchell MN, Culver N, Kay M, McGowan SK, Song Y, Deleeuw C, Martin JL. Values Expressed by Women Veterans Receiving Treatment for Chronic Insomnia Disorder. Behav Sleep Med. 2024 May-Jun;22(3):340-352. doi: 10.1080/15402002.2023.2260517. Epub 2023 Sep 25. PMID 37749876
- [Derived] Martin JL, Carlson GC, Kelly MR, Song Y, Mitchell MN, Josephson KR, McGowan SK, Culver NC, Kay MA, Erickson AJ, Saldana KS, May KJ, Fiorentino L, Alessi CA, Washington DL, Yano EM. Novel treatment based on acceptance and commitment therapy versus cognitive behavioral therapy for insomnia: A randomized comparative effectiveness trial in women veterans. J Consult Clin Psychol. 2023 Nov;91(11):626-639. doi: 10.1037/ccp0000836. Epub 2023 Aug 3. PMID 37535521
- [Derived] Carlson GC, Kelly MR, Grinberg AM, Mitchell M, McGowan SK, Culver NC, Kay M, Alessi CA, Washington DL, Yano EM, Martin JL. Insomnia Precipitating Events among Women Veterans: The Impact of Traumatic and Nontraumatic Events on Sleep and Mental Health Symptoms. Behav Sleep Med. 2021 Sep-Oct;19(5):672-688. doi: 10.1080/15402002.2020.1846537. Epub 2020 Nov 30. PMID 33251855

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 347 subjects were enrolled into the study (i.e., signed consent) and were administered the baseline assessment. Final eligibility determination was made after baseline assessments. Only participants who met final inclusion/exclusion criteria (after baseline) were eligible for randomization. Results are only provided for the 149 randomized subjects.
Groups:
- ABC-I: Experimental: ABC-I Participants completed a 5 session intervention, Acceptance and the Behavioral Changes to Treat Insomnia (ABC-I). This was considered the "new treatment" being studied.
- CBT-I: Active Comparator: CBT-I Participants received a 5-session intervention, cognitive-behavioral therapy for insomnia (CBT-I). This was considered the "standard care" treatment.
Period: Overall Study
Arm/Group | ABC-I | CBT-I
Started | 74 | 75
Completed | 66 | 69
Not Completed | 8 | 6
Not completed — Lost to Follow-up | 7 | 5
Not completed — Refused follow-up assessment | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- ABC-I: Participants will participate in 5 individual sessions with a trained instructor.
  Behavioral treatment for insomnia-Group I: Participants will attend 5 individual sessions with a trained instructor.
- CBT-I: Participants will participate in 5 individual sessions with a trained instructor.
  Behavioral treatment for insomnia-Group II: Participants will attend in 5 individual sessions with a trained instructor.
- Total: Total of all reporting groups
Arm/Group | ABC-I | CBT-I | Total
Number analyzed (Participants) | 74 | 75 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.89 (12.68) | 47.76 (13.53) | 47.82 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 75 | 149
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 17 | 34
  Not Hispanic or Latino | 57 | 58 | 115
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 27 | 41
  White | 40 | 41 | 81
  More than one race | 10 | 5 | 15
  Unknown or Not Reported | 5 | 1 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 74 | 75 | 149
Insomnia Severity Index (ISI) [Mean (Standard Deviation); unit: units on a scale] — The Insomnia Severity Index (ISI) is a 7-item scale instrument that measures perceived severity of insomnia symptoms. Score ranges from 0 to 28, with higher scores indicating greater insomnia severity.
  units on a scale | 14.19 (4.82) | 14.57 (5.12) | 14.38 (4.96)
Patient Health Questionnaire-9 (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — The PHQ-9 is a 9-item depression module in the Patient Health Questionnaire (a self-administered diagnostic instrument for common mental disorders) which is part of the Primary Care Evaluation of Mental Disorders (PRIME-MD) suite of evaluation tools. Scores range from 0 to 27 with higher scores indicating greater depression symptom severity.
  units on a scale | 10.55 (5.67) | 10.28 (5.42) | 10.42 (5.53)
PTSD Checklist for DSM-5 [Mean (Standard Deviation); unit: units on a scale] — The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure that assesses the presence and severity of PTSD symptoms. Items on the PCL-5 correspond with DSM-5 criteria for PTSD. Scores range from 0 to 80 with higher scores indicating greater severity of PTSD symptoms.
  units on a scale | 26.25 (21.81) | 25.28 (20.97) | 25.75 (21.32)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Completing 5 Behavioral Treatment Sessions
Description: Number of participants who attended and completed all 5 behavioral treatment sessions.
Time Frame: End of the 5-week behavioral treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | ABC-I | CBT-I
Number analyzed (Participants) | 74 | 75
Participants | 63 | 70
Statistical Analysis 1: Comparison: ABC-I vs CBT-I; Percentage of participants who completed all 5 treatment sessions, comparing ABC-I to CBT-I; Test type: Superiority; p = .120, Fisher Exact

2. Primary Outcome: Adherence With Bedtime Recommendations
Description: Minutes deviation from recommended bedtime recommendations during final week of intervention period.
Time Frame: Final 7 nights of the 5-week intervention period
Measure: Mean (Standard Error); unit: minutes
Arm/Group | ABC-I | CBT-I
Number analyzed (Participants) | 74 | 75
minutes | -6.43 (2.59) | -5.71 (2.48)
Statistical Analysis 1: Comparison: ABC-I vs CBT-I; Test type: Superiority; p = .843, Mixed Models Analysis; Mean Difference (Final Values) = -.711, 95% CI 2-sided [-7.75 to 6.32], Standard Error of Mean 3.59 — The average deviation, in minutes, between the recommended and actual bed time. Negative values indicate the number of minutes earlier than the recommended bed time that the participant went to bed, indicating greater non-adherence

3. Primary Outcome: Adherence to Rise Time Recommendations
Description: Minutes deviation from recommended rise time during the final week of the intervention period
Time Frame: Final 7-nights of the 5-week intervention period
Measure: Mean (Standard Error); unit: minutes
Arm/Group | ABC-I | CBT-I
Number analyzed (Participants) | 74 | 75
minutes | 20.63 (3.73) | 23.41 (3.58)
Statistical Analysis 1: Comparison: ABC-I vs CBT-I; Test type: Superiority; p = 0.590, Mixed Models Analysis; Mean Difference (Final Values) = -2.78, 95% CI 2-sided [-12.91 to 7.35], Standard Error of Mean 5.17 — The average deviation, in minutes, between the recommended and actual rise time. Positive values indicate the number of minutes later than the recommended rise time that the participant got out of bed, indicating greater non-adherence

4. Primary Outcome: Non-adherence to Nighttime Stimulus Control
Description: Average proportion of nights on which participant did not get out of bed if unable to sleep after 20 minutes awake.
Time Frame: Final 7-nights of the 5-week intervention period
Measure: Mean (Standard Error); unit: Proportion of nights
Arm/Group | ABC-I | CBT-I
Number analyzed (Participants) | 74 | 75
Proportion of nights | .274 (.035) | .273 (.033)
Statistical Analysis 1: Comparison: ABC-I vs CBT-I; Test type: Superiority; p = 0.979, Mixed Models Analysis; Mean Difference (Final Values) = .001, 95% CI 2-sided [-0.093 to 0.096], Standard Error of Mean 0.048 — The proportion of nights participants who did not follow the recommendation to get out of bed if awake more than 20 minutes. Higher numbers indicate greater non-adherence

5. Secondary Outcome: Sleep Efficiency From Sleep Diary at Post-Treatment
Description: Sleep efficiency (mean percent time asleep while in bed) will be calculated from 7 days of self-reported sleep diary.
Time Frame: 1 week after the end of the 5-week intervention period
Measure: Mean (Standard Error); unit: percentage of time asleep
Arm/Group | ABC-I | CBT-I
Number analyzed (Participants) | 74 | 75
percentage of time asleep | 13.88 (1.45) | 13.47 (1.41)
Statistical Analysis 1: Comparison: ABC-I vs CBT-I; Test type: Non-Inferiority — We elected to use a value of δ equivalent to an effect size of d=0.40. (i.e., 4/10ths SD). For sleep diary estimated sleep efficiency, this represents a difference of 5%; p = 0.004, Mixed Models Analysis; Mean Difference (Net) = 0.409, 90% CI 2-sided [-2.92 to 3.74], Standard Error of Mean 2.02 — The parameter estimate is the improvement in sleep efficiency from baseline to post-treatment for ABCI group versus the same improvement in the CBTI group

6. Secondary Outcome: Sleep Efficiency From Sleep Diary at 3-month Follow-up
Description: Sleep efficiency (mean percent time asleep while in bed) will be calculated from 7 days of self-reported sleep diary.
Time Frame: 3-months after randomization
Measure: Mean (Standard Error); unit: percentage of time asleep
Arm/Group | ABC-I | CBT-I
Number analyzed (Participants) | 74 | 75
percentage of time asleep | 12.74 (1.52) | 11.98 (1.47)
Statistical Analysis 1: Comparison: ABC-I vs CBT-I; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p = .003, Mixed Models Analysis; Mean Difference (Net) = 0.757, 90% CI 2-sided [-2.72 to 4.23], Standard Error of Mean 2.12 — The parameter estimate is the improvement in sleep efficiency from baseline to 3-month follow-up for ABCI group versus the same improvement in the CBTI group

7. Secondary Outcome: Sleep Efficiency From Actigraphy at Post-Treatment
Description: Sleep efficiency (mean percent time asleep while in bed) will be calculated from 7 days of wrist actigraphy.
Time Frame: 1 week after the end of the 5-week intervention period
Measure: Mean (Standard Error); unit: percentage of time asleep
Arm/Group | ABC-I | CBT-I
Number analyzed (Participants) | 74 | 75
percentage of time asleep | 2.32 (0.83) | 1.64 (0.79)
Statistical Analysis 1: Comparison: ABC-I vs CBT-I; Test type: Non-Inferiority — We elected to use a value of δ equivalent to an effect size of d=0.40. (i.e., 4/10ths SD). For actigraphically-estimated sleep efficiency, this represents a difference of 5%; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 0.68, 90% CI 2-sided [-1.21 to 2.57], Standard Error of Mean 1.15 — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: Sleep Efficiency From Wrist Actigraphy at 3-month Follow-up
Description: Sleep efficiency (mean percent time asleep while in bed) will be calculated from 7 days of wrist actigraphy.
Time Frame: 3-months after randomization
Measure: Mean (Standard Error); unit: percentage of time asleep
Arm/Group | ABC-I | CBT-I
Number analyzed (Participants) | 74 | 75
percentage of time asleep | 1.33 (0.99) | 0.22 (0.94)
Statistical Analysis 1: Comparison: ABC-I vs CBT-I; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < .001, Mixed Models Analysis; Mean Difference (Net) = 1.11, 90% CI 2-sided [-1.14 to 3.36], Standard Error of Mean 1.37 — [estimate comment as in outcome 6, analysis 1]

9. Secondary Outcome: Change From Baseline to Post-Treatment in Insomnia Severity Index Score
Description: Mean score on Insomnia Severity Index (ISI). This 7-item scale measures self-reported severity of insomnia symptoms. Total score ranges from 0 to 28, with higher scores indicating greater insomnia severity.
Time Frame: Baseline and 1 week after the end of the 5-week intervention period
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ABC-I | CBT-I
Number analyzed (Participants) | 74 | 75
score on a scale | -8.68 (0.65) | -9.18 (0.62)
Statistical Analysis 1: Comparison: ABC-I vs CBT-I; Test type: Non-Inferiority — We elected to use a value of δ equivalent to an effect size of d=0.40. (i.e., 4/10ths SD). With respect to ISI, this represents a 2 point difference between the treatment effects; p = 0.048, Mixed Models Analysis; Mean Difference (Net) = 0.501, 90% CI 2-sided [-0.98 to 1.98], Standard Error of Mean 0.90 — The parameter estimate is the improvement in the ISI score from baseline to post-treatment for ABCI group versus the same improvement in the CBTI group

10. Secondary Outcome: Change From Baseline to 3-month Follow-up in Insomnia Severity Index Score
Description: as for outcome 9
Time Frame: Baseline and 3-months from randomization
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ABC-I | CBT-I
Number analyzed (Participants) | 74 | 75
score on a scale | -8.29 (0.76) | -7.71 (0.74)
Statistical Analysis 1: Comparison: ABC-I vs CBT-I; Test type: Non-Inferiority — [test comment as in outcome 9, analysis 1]; p = 0.008, Mixed Models Analysis; Mean Difference (Net) = -0.57, 90% CI 2-sided [-2.32 to 1.17], Standard Error of Mean 1.06 — The parameter estimate is the improvement in the ISI score from baseline to 3-month follow-up for ABCI group versus the same improvement in the CBTI group

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 3 months.
Arm/Group | ABC-I | CBT-I
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/75
Other Adverse Events (participants affected / at risk) | 0/74 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2016-08-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT02076165/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/65/NCT02076165/Prot_SAP_001.pdf